CLINICAL TRIAL: NCT02678221
Title: Sildenafil Citrate for the Management of Asymmetrical Intrauterine Growth Restriction
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Mamdouh Shaaban, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SCIUGR
Record Dates: First submitted 2016-02-05; First posted 2016-02-09 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Intrauterine Growth Restriction
MeSH Terms: conditions — Fetal Growth Retardation | interventions — Sildenafil Citrate; Aspirin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sildenafil citrate with Aspirin (Active Comparator): will receive sildenafil citrate 20mg ̸ 8hours plus low dose aspirin 150mg/day
  Interventions: Drug: Sildenafil citrate; Drug: Aspirin
- placebo with Aspirin (Other): will receive placebo plus low dose aspirin 150mg/day
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Sildenafil citrate
  Arms: Sildenafil citrate with Aspirin
Drug: Aspirin

SUMMARY:
Intrauterine growth restriction (IUGR) is defined as fetal abdominal circumference (AC) or estimated fetal weight (EFW) < 10th centile. In asymmetrical IUGR the parameter classically affected is the abdominal circumference (AC). Fetal growth restriction (FGR) complicates approximately 0.4% of pregnancies and severely increases the risk of perinatal morbidity and mortality. This is particularly due to premature delivery, both for fetal and for secondary maternal indications such as the development of pre-eclampsia.

Consequence of deficient uteroplacental blood flow, including IUGR, pre-eclampsia, and placental abruption have been implicated in more than 50% of iatrogenic premature births. For this reason, the problem of severe IUGR forms a substantial portion of the population that tertiary care centres care for.

The effect of early-onset IUGR is particularly significant: of those born alive, less than a third will survive their neonatal intensive care unit (NICU) stay without significant neurodevelopmental sequelae. Survival rates for severely growth-restricted fetuses very remote from term (<28 weeks' gestation) vary from 7% to 33%.

As these early-onset IUGR children are born very preterm, there are significant risks of neonatal mortality, major and minor morbidity, and long-term health sequelae.

The use of ultrasound Doppler waveform analysis in pregnancies complicated by IUGR suggests compromised uteroplacental circulation and placental hypoperfusion. Currently there are no specific evidence-based therapies for placental insufficiency and severe IUGR. Non-specific interventions include primarily lifestyle modifications, such as reducing or stopping work, stopping aerobic exercise, rest at home, and hospital admission for rest and surveillance. These interventions, which are not supported by evidence from randomized trials, are used in the belief that rest will enhance the uteroplacental circulation at the expense of that to the glutei and quadriceps muscles.

There is evidence from ex vivo and animal models of growth restriction that the phosphodiesterase 5 inhibitor sildenafil citrate increases average birth weight and improves uteroplacental blood flow (umbilical artery, uterine artery).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant Women ≥ 28 wk
* Diagnosed as asymmetrical Intrauterine growth restriction

Exclusion Criteria:

* Severe preeclampsia
* Fetus with reversed umbilical artery end diastolic flow.
* Symmetrical Intrauterine growth restriction
* Diagnosed to have congenital anomalies.
* Diabetes mellitus with pregnancy.
* Patients with contraindication for the drugs given as gastric or duodenal ulcer,
* Twins pregnancy.
* Patients on antihypertensive or rheumatic heart disease
* Smokers.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-02 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
The fetal weight by grams | 1 year

SECONDARY OUTCOMES:
Doppler indices changes in umbilical artery and middle cerebral artery. | 1 year
Maternal blood pressure changes. | 1 year
Number of babies admitted to Pediatric Care Unit. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Asyut, Asyut Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes